CLINICAL TRIAL: NCT04646629
Title: Effect of Electroacupuncture on Sepsis-induced Intestinal Dysfunction: a Prospective, Double-blind, Randomized Controlled Trial
Brief Title: Effect of Electroacupuncture on Sepsis-induced Intestinal Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jianbo Yu (Other)
Responsible Party: Sponsor-Investigator, Jianbo Yu, Department of Anesthesiology, Director, Chief physician, Professor, Doctoral tutor, Tianjin Nankai Hospital
Organization: Tianjin Nankai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKYY_YXKT_IRB_2020_071_01
Record Dates: First submitted 2020-11-22; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Sepsis; Intestinal Dysfunction
Keywords: sepsis; electroacupuncture; intestinal dysfunction
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture treatment (Experimental): Participants in the treatment group underwent 60 minutes acupuncture (0.30mm×70mm) at ST36 (Zusanli) and ST37 (Shangjuxu) twice a day for seven days. After"Deqi",electroacupuncture stimulation apparatus (HANS G6805-2, Huayi Co, Shanghai, China) isconnected and maintained the end of treatment
  Interventions: Device: electroacupuncture treatment
- sham electroacupuncture treatment (Sham Comparator): sham electroacupuncture treatment participants in the control group received shallow needling (0.30mm×25mm) at ST36 and ST37(nonacupoints located 1 inch beside acupoints, about 20mm). Specifically, the depth of needle insertion into nonacupoints is 3-5mm and avoided manual stimulation and no "Deqi" without actual current output.
  Interventions: Device: sham electroacupuncture treatment

INTERVENTIONS:
Device: electroacupuncture treatment — Participants in the treatment group underwent 60 minutes acupuncture (0.30mm×70mm) at ST36 (Zusanli) and ST37 (Shangjuxu) twice a day for seven days.After "Deqi", electroacupuncture stimulation apparatus (HANS G6805-2, Huayi Co, Shanghai, China) is connected with the density wave (2/100 Hz), width 0.25 ms, intensity of 1 ~ 30 mA (gradually increase to the patient's maximum tolerance) and maintained the end of treatment.
  Arms: electroacupuncture treatment
Device: sham electroacupuncture treatment — Participants in the sham electroacupuncture group received shallow needling (0.30mm×25mm) at ST36 and ST37(nonacupoints located 1 inch beside acupoints, about20mm). Specifically, the depth of needle insertion into nonacupoints is 3-5mm and avoided manual stimulation and no "Deqi" without actual current output, and retained the needle for the same time as treatment group
  Arms: sham electroacupuncture treatment

SUMMARY:
1. Title: Effect of electroacupuncture on sepsis-induced intestinal dysfunction
2. Research center: single center
3. The Design of the study: Randomized, double-blind, controlled study
4. The population of the study: The patients over 18 years that met the criteria of sepsis3.0 and with AGI grade II or above are enrolled in the study
5. Sample size: Enroll 60 patients (30patients in each group)
6. Interventions: Participants in the treatment group underwent 60 minutes acupuncture (0.30mm×70mm) at ST36 (Zusanli) and ST37 (Shangjuxu) twice a day for seven days. After"Deqi",electroacupuncture stimulation apparatus (HANS G6805-2, Huayi Co, Shanghai, China) is connected and maintained the end of treatment.

   Participants in the control group received shallow needling (0.30mm×25mm) at ST36 and ST37(nonacupoints located 1 inch beside acupoints, about 20mm). Specifically, the depth of needle insertion into nonacupoints is 3-5mm and avoided manual stimulation and no "Deqi" without actual current output.
7. The aim of the research: To investigate the effect of electroacupuncture on sepsis-induced intestinal dysfunction.
8. Outcome# 1) Primary outcome: The intestinal function indicators including: 1) Clinical symptoms: bowel sounds, intra-abdominal pressure, time to first exhaust/defecation, daily tolerable enteral nutrition 2) Intestinal motility indicators: the levels of serum motilin and gastrin 3) Intestinal barrier indicators: the levels of serum diamine oxidase (DAO), D-lactic acid and I-FABP 2)Secondary outcome# Duration of mechanical ventilation in patients with endotracheal intubation on ICU admission; Length of stay in ICU and Length of stay in hospital; 30-day life quality and cognitive function after surgery; All-cause 28-day mortality.
9. The estimated duration of the study#1-2years.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, placebo controlled and long-term follow-up design. In this study, ST36 (Zusanli) and ST37 (Shangjuxu) were selected for electroacupuncture treatment, accompanied with evaluating the effects on intestinal function in septic patients. Meanwhile, the blood biochemical indexes such as heme oxygenase-1(HO-1), PTEN induced putative kinase 1(PINK1), polo-like kinase 1(PLK1) and interleukin-6 are detected. To clarify the effect of electroacupuncture on sepsis-induced intestinal dysfunction is of great significance to the clinical applications and popularization of traditional acupuncture treatment across the world.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of sepsis 3.0
2. AGI grade II or above,
3. At least 18 years old
4. Volunteer to participate in this study and sign the informed consent form

Exclusion Criteria:

1. Patients with bowel dysfunction caused by other diseases or surgical operations
2. Those who have chronic gastrointestinal diseases such as Crohn's disease and ulcerative colitis
3. Those who have recently used gastrointestinal motility drugs and within 5 times the half-life
4. Those who are participating in other drug clinical trials
5. Refuse to participate in this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-23 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The effect on intestinal motility | an average of one year
  Record the serum levels of motilin of the two groups
The effect on intestinal motility | an average of 1 year
  Record the serum levels of gastrin of the two groups
The effect on intestinal barrier | up to 1 year
  Record serum levels of DAO of the two groups
The effect on intestinal barrier | up to 12 months
  Record serum levels of I-FABP of the two groups

SECONDARY OUTCOMES:
Duration of mechanical ventilation in patients with endotracheal intubation in ICU | one year
  Duration of mechanical ventilation and endotracheal intubation in ICU
Length of stay in hospital | up to one year
  ICU stay time and hospitalization time
All-cause 28-day mortality | 12 months
  All reasons (such as infection, hemorrhage) caused the mortality during the first 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Yu, PhD, Study Chair — Tianjin Nankai Hospital
Locations (1):
- Electroacupuncture Apparatus, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meng JB, Jiao YN, Zhang G, Xu XJ, Ji CL, Hu MH, Lai ZZ, Zhang M. Electroacupuncture Improves Intestinal Dysfunction in Septic Patients: A Randomised Controlled Trial. Biomed Res Int. 2018 Jun 26;2018:8293594. doi: 10.1155/2018/8293594. eCollection 2018. PMID 30046610
- [Background] Yoseph BP, Klingensmith NJ, Liang Z, Breed ER, Burd EM, Mittal R, Dominguez JA, Petrie B, Ford ML, Coopersmith CM. Mechanisms of Intestinal Barrier Dysfunction in Sepsis. Shock. 2016 Jul;46(1):52-9. doi: 10.1097/SHK.0000000000000565. PMID 27299587
- [Background] Li HF, Hu GQ, Liu WW. [Clinical trials of acupuncture of Jiaji (EX-B2) for treatment of gastrointestinal dysfunction in sepsis patients]. Zhen Ci Yan Jiu. 2019 Jan 25;44(1):43-6. doi: 10.13702/j.1000-0607.170579. Chinese. PMID 30773861
- [Background] Liu H, Zhu J, Ni HB, Hu XX. [Transcutaneous electrical acupoint stimulation for early enteral nutrition tolerance in patients with sepsis of gastrointestinal dysfunction: a multi-center randomized controlled trial]. Zhongguo Zhen Jiu. 2020 Mar 12;40(3):229-33. doi: 10.13703/j.0255-2930.20190426-0003. Chinese. PMID 32270631